CLINICAL TRIAL: NCT00295022
Title: Double-blind, Three Parallel Randomized Groups, Therapeutic Confirmatory Clinical Trial to Compare the Efficacy of Oral Levocetirizine 5 mg and Montelukast 10 mg to Placebo in Reducing Symptoms of Seasonal Allergic Rhinitis (SAR) in Ragweed Sensitive Subjects Exposed to Ragweed Pollen in an Environmental Exposure Unit (EEU)
Brief Title: Compare the Efficacy of Levocetirizine and Montelukast to Placebo in Reducing Seasonal Allergic Rhinitis (SAR) Symptoms in Ragweed Sensitive Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB S.A. - Pharma Sector (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A00414
Record Dates: First submitted 2006-02-20; First posted 2006-02-22 (Estimated); Results first posted 2018-07-23 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: Levocetirizine; Xyzal; Rhinitis; Allergic; Seasonal; Ragweed
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis | interventions — montelukast; levocetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (PBO) (Placebo Comparator): Placebo was administered orally on Days 1 and 2.
  Interventions: Drug: Placebo
- Montelukast (MLKT) (Experimental): 10 mg of Montelukast (MLKT) was administered orally on Days 1 and 2.
  Interventions: Drug: Montelukast
- Levocetirizine (LCTZ) (Experimental): 5 mg of Levocetirizine (LCTZ) was administered orally on Days 1 and 2.
  Interventions: Drug: Levocetirizine

INTERVENTIONS:
Drug: Placebo — * Pharmaceutical form: Over-encapsulated tablet
  * Route of administration: Oral use
  Arms: Placebo (PBO)
Drug: Montelukast — * Pharmaceutical form: Over-encapsulated tablet
  * Concentration: 10 mg
  * Route of administration: Oral use
  Arms: Montelukast (MLKT)
Drug: Levocetirizine — * Pharmaceutical form: Over-encapsulated tablet
  * Concentration: 5 mg
  * Route of administration: Oral use
  Arms: Levocetirizine (LCTZ)

SUMMARY:
To compare the clinical efficacy of levocetirizine 5 mg and montelukast 10 mg on symptoms of seasonal allergic rhinitis occurring in subjects exposed to ragweed pollen in an environmental exposure unit.

ELIGIBILITY:
Inclusion Criteria:

* Have had seasonal allergic rhinitis due to Ragweed for the last 2 consecutive years
* Subjects who obtain a minimum sum score, considering Seasonal Allergic Rhinitis (SAR) related symptoms (mean value), as defined by the protocol

Exclusion Criteria:

* Any clinically significant condition that might interfere with the treatment evaluation, both for efficacy and safety
* Have used forbidden concomitant medications as defined by the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2006-07-29; Primary Completion 2006-10-01 (Actual); Study Completion 2006-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — UCB (+1 844 599 2273)
Locations (1):
- Kingston, Ontario, Canada

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant Flow refers to the Randomized Set.
Period: Overall Study
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) | Montelukast (MLKT)
Started | 105 | 157 | 156
Completed | 104 | 156 | 151
Not Completed | 1 | 1 | 5
Not completed — Adverse Event | 1 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Intention-To-Treat (ITT) Set
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) | Montelukast (MLKT) | Total Title
Number analyzed (Participants) | 105 | 157 | 156 | 418
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 104 | 155 | 156 | 415
  >=65 years | 1 | 2 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.41 (11.74) | 34.95 (11.98) | 32.98 (11.72) | 34.33 (11.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 101 | 89 | 250
  Male | 45 | 56 | 67 | 168

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Major Symptom Complex (MSC) Score Over Period I
Description: Six individual symptoms which are most dominant in the rhinitis symptom profile will be combined to form the MSC severity score:
  Runny nose (right and left), itchy nose (right and left), sniffles, nose blows, sneezes, watery eyes.
  Each individual symptom, except nose blows and sneezes, is rated on a 5-point scale of severity: 0 = None, 1 = a little, 2 = Moderate, 3 = Quite a bit, 4 = severe, 5 = very severe. For nose blows and sneezes, the subjects had to record the number of each symptom since last evaluation. This number corresponds to a score ranging from 0 to 8. The total MSC score ranges from 0 - 36. Increasing scores are associated with increasing severity. Negative values indicate improvement from Baseline.
Time Frame: Baseline, Treatment Period 1 [Day 1, from drug intake (at 11:00 am) to 5 hours post-treatment (at 4:00 pm)]
Population: Efficacy variables were analyzed using the Intention-To-Treat (ITT) population. ITT consists of all randomized subjects who took at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) | Montelukast (MLKT)
Number analyzed (Participants) | 105 | 157 | 156
units on a scale | -3.46 (0.49) | -6.58 (0.40) | -5.65 (0.40)
Statistical Analysis 1: Comparison: Placebo (PBO) vs Levocetirizine (LCTZ); Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -3.12, 95% CI 2-sided [-4.35 to -1.88]
Statistical Analysis 2: Comparison: Levocetirizine (LCTZ) vs Montelukast (MLKT); Test type: Superiority or Other; p = 0.001, ANCOVA; Mean Difference (Final Values) = -0.93, 95% CI 2-sided [-2.04 to 0.18]
Statistical Analysis 3: Comparison: Placebo (PBO) vs Montelukast (MLKT); Test type: Superiority or Other; p < 0.001, ANCOVA; Median Difference (Final Values) = -2.19, 95% CI 2-sided [-3.43 to -0.95]

2. Secondary Outcome: Change From Baseline in the MSC Score Over Period II
Description: as for outcome 1
Time Frame: Baseline, Treatment Period II [Day 2, from 9:30 am to 11:00 am]
Population: Only patients with valid MSC scores in Period II were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) | Montelukast (MLKT)
Number analyzed (Participants) | 104 | 156 | 151
units on a scale | -1.22 (0.52) | -6.35 (0.42) | -3.24 (0.43)

3. Secondary Outcome: Change From Baseline in the MSC Score Over Period III
Description: as for outcome 1
Time Frame: Baseline, Treatment Period III [Day 2, from drug intake (at 11:00 am) to 3:30 pm]
Population: Only patients with valid MSC scores in Period III were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Montelukast (MLKT) | Levocetirizine (LCTZ)
Number analyzed (Participants) | 104 | 151 | 156
units on a scale | -3.50 (0.58) | -8.62 (0.47) | -6.19 (0.48)

4. Secondary Outcome: Change From Baseline in the MSC Score Over the Total Treatment Period (Period I + Period II + Period III)
Description: as for outcome 1
Time Frame: Baseline to Day 2
Population: Only patients with valid MSC scores during the Total Treatment Period were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) | Montelukast (MLKT)
Number analyzed (Participants) | 105 | 157 | 156
units on a scale | -3.16 (0.46) | -7.37 (0.38) | -5.48 (0.38)

5. Secondary Outcome: Change From Baseline in the Total Symptom Complex (TSC) Score Over Period I
Description: The TSC score was calculated as the sum of the following 10 individual symptom scores:
  runny nose (left and right), itchy nose (left and right), sniffles, nose blows, sneezes, watery eyes, itchy eyes and ears, itchy throat, cough and postnasal drip.
  Each individual symptom, except nose blows and sneezes, is rated on a 5-point scale of severity: 0 = None, 1 = a little, 2 = Moderate, 3 = Quite a bit, 4 = severe, 5 = very severe. For nose blows and sneezes, the subjects had to record the number of each symptom since last evaluation. This number corresponds to a score ranging from 0 to 8. The TSC score ranges from 0 to 56. Increasing scores are associated with increasing severity. Negative values indicate improvement from Baseline.
Time Frame: Baseline, Treatment Period 1 [Day 1, from drug intake (at 11:00 am) to 5 hours post-treatment (at 4:00 pm)]
Population: Only patients with valid TSC scores in Period I were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) | Montelukast (MLKT)
Number analyzed (Participants) | 105 | 157 | 156
units on a scale | -6.16 (0.75) | -10.53 (0.61) | -9.01 (0.61)

6. Secondary Outcome: Change From Baseline in the Total Symptom Complex (TSC) Score Over Period II
Description: as for outcome 5
Time Frame: Baseline, Treatment Period II [Day 2, from 9:30 am to 11:00 am]
Population: Only patients with valid TSC scores in Period II were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) | Montelukast (MLKT)
Number analyzed (Participants) | 104 | 156 | 151
units on a scale | -2.45 (0.76) | -9.54 (0.62) | -5.12 (0.63)

7. Secondary Outcome: Change From Baseline in the Total Symptom Complex (TSC) Score Over Period III
Description: as for outcome 5
Time Frame: Baseline, Treatment Period III [Day 2, from drug intake (at 11:00 am) to 3:30 pm]
Population: Only patients with valid TSC scores in Period III were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) | Montelukast (MLKT)
Number analyzed (Participants) | 104 | 156 | 151
units on a scale | -5.91 (0.88) | -13.39 (0.72) | -9.73 (0.73)

8. Secondary Outcome: Change From Baseline in the Total Symptom Complex (TSC) Score Over the Total Treatment Period (Period I + Period II + Period III)
Description: as for outcome 5
Time Frame: Baseline to Day 2
Population: Only patients with valid TSC scores during the Total Treatment Period were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) | Montelukast (MLKT)
Number analyzed (Participants) | 105 | 157 | 156
units on a scale | -5.53 (0.72) | -11.54 (0.59) | -8.68 (0.59)

9. Secondary Outcome: Change From Baseline in the TSC Score + Nasal Congestion Score Over Period I
Description: The TSC score was calculated as the sum of the following 10 individual symptom scores:
  runny nose (left and right), itchy nose (left and right), sniffles, nose blows, sneezes, watery eyes, itchy eyes and ears, itchy throat, cough and postnasal drip.
  Each individual symptom, except nose blows and sneezes, is rated on a 5-point scale of severity: 0 = None, 1 = a little, 2 = Moderate, 3 = Quite a bit, 4 = severe, 5 = very severe. For nose blows and sneezes, the subjects had to record the number of each symptom since last evaluation. This number corresponds to a score ranging from 0 to 8.
  The Nasal congestion score ranged from 0 to 4 (0 = clear, 1 = slight block, 2 = stuffy, 3 = very stuffy, 4 = blocked). It corresponds to the mean value of right nostril and left nostril. The TSC score plus Nasal congestion score was added and ranged from 0 to 60. Increasing scores are associated with increasing severity. Negative values indicate improvement from Baseline.
Time Frame: Baseline, Treatment Period 1 [Day 1, from drug intake (at 11:00 am) to 5 hours post-treatment (at 4:00 pm)]
Population: Only patients with valid TSC score + Nasal congestion score in Period I were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) | Montelukast (MLKT)
Number analyzed (Participants) | 105 | 157 | 156
units on a scale | -6.57 (0.80) | -11.15 (0.66) | -9.65 (0.66)

10. Secondary Outcome: Change From Baseline in the TSC Score + Nasal Congestion Score Over Period II
Description: as for outcome 9
Time Frame: Baseline, Treatment Period II [Day 2, from 9:30 am to 11:00 am]
Population: Only patients with valid TSC score + Nasal congestion score in Period II were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) | Montelukast (MLKT)
Number analyzed (Participants) | 104 | 156 | 151
units on a scale | -2.65 (0.80) | -9.97 (0.65) | -5.47 (0.66)

11. Secondary Outcome: Change From Baseline in the TSC Score + Nasal Congestion Score Over Period III
Description: as for outcome 9
Time Frame: Baseline, Treatment Period III [Day 2, from drug intake (at 11:00 am) to 3:30 pm]
Population: Only patients with valid TSC score + Nasal congestion score in Period III were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) | Montelukast (MLKT)
Number analyzed (Participants) | 104 | 156 | 151
units on a scale | -6.35 (0.94) | -14.18 (0.77) | -10.39 (0.78)

12. Secondary Outcome: Change From Baseline in the TSC Score + Nasal Congestion Score Over the Total Treatment Period (Period I + Period II + Period III)
Description: as for outcome 9
Time Frame: Baseline to Day 2
Population: Only patients with valid TSC score + Nasal congestion score during the Total Treatment Period were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) | Montelukast (MLKT)
Number analyzed (Participants) | 105 | 157 | 156
units on a scale | -5.92 (0.77) | -12.21 (0.63) | -9.28 (0.63)

13. Secondary Outcome: Change From Baseline in the Individual Symptom Scores Over Period I
Description: Individual symptom scores include Runny Nose Score, Itchy Nose Score, Sniffles Score, Postnasal Drip Score, Watery Eyes Score, Itchy Eyes and Ears Score, Itchy Throat Score, Cough Score, Sneezes Score, Nose Blows Score, Nasal Congestion Score.
  The subjects had to evaluate the severity of the symptoms using a scale from "None" to "Very severe" (ranging from 0 to 5).
  For Sneezes Score and Nose Blows Score, the subjects had to record the number of each symptom since last evaluation. This number corresponds to a score ranging from 0 to 8.
  The Nasal congestion score ranged from 0 to 4 (0 = clear, 1 = slight block, 2 = stuffy, 3 = very stuffy, 4 = blocked). It corresponds to the mean value of right nostril and left nostril.
  Increasing scores are associated with increasing severity. Negative values indicate improvement from Baseline.
Time Frame: Baseline, Treatment Period 1 [Day 1, from drug intake (at 11:00 am) to 5 hours post-treatment (at 4:00 pm)]
Population: Only patients with valid individual symptom scores in Period I were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) | Montelukast (MLKT)
Number analyzed (Participants) | 105 | 157 | 156
units on a scale
  Runny Nose Score | -0.55 (0.09) | -0.89 (0.07) | -0.86 (0.07)
  Itchy Nose Score | -0.52 (0.09) | -0.93 (0.08) | -0.85 (0.08)
  Sniffles Score | -0.53 (0.09) | -0.93 (0.08) | -0.87 (0.08)
  Postnasal Drip Score | -0.65 (0.10) | -0.99 (0.08) | -0.89 (0.08)
  Watery Eyes Score | -0.58 (0.09) | -0.94 (0.07) | -0.82 (0.07)
  Itchy Eyes/Ears Score | -0.69 (0.09) | -1.14 (0.08) | -0.90 (0.08)
  Itchy Throat Score | -0.66 (0.09) | -1.00 (0.07) | -0.85 (0.07)
  Cough Score | -0.71 (0.06) | -0.81 (0.05) | -0.71 (0.05)
  Sneezes Score | -0.28 (0.11) | -1.07 (0.09) | -0.68 (0.09)
  Nose Blows Score | -1.03 (0.13) | -1.77 (0.10) | -1.59 (0.10)
  Nasal Congestion Score | -0.41 (0.07) | -0.62 (0.06) | -0.64 (0.06)

14. Secondary Outcome: Change From Baseline in the Individual Symptom Scores Over Period II
Description: as for outcome 13
Time Frame: Baseline, Treatment Period II [Day 2, from 9:30 am to 11:00 am]
Population: Only patients with valid individual symptom scores in Period II were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) | Montelukast (MLKT)
Number analyzed (Participants) | 104 | 156 | 151
units on a scale
  Runny Nose Score | -0.18 (0.09) | -0.85 (0.08) | -0.53 (0.08)
  Itchy Nose Score | -0.22 (0.09) | -0.84 (0.07) | -0.40 (0.08)
  Sniffles Score | -0.10 (0.09) | -0.83 (0.08) | -0.48 (0.08)
  Postnasal Drip Score | -0.37 (0.09) | -0.90 (0.08) | -0.52 (0.08)
  Watery Eyes Score | -0.20 (0.11) | -0.66 (0.09) | -0.46 (0.09)
  Itchy Eyes/Ears Score | -0.18 (0.10) | -0.81 (0.08) | -0.40 (0.09)
  Itchy Throat Score | -0.19 (0.10) | -0.78 (0.08) | -0.39 (0.09)
  Cough Score | -0.49 (0.08) | -0.70 (0.06) | -0.58 (0.06)
  Sneezes Score | -0.19 (0.14) | -1.28 (0.11) | -0.40 (0.12)
  Nose Blows Score | -0.38 (0.15) | -1.84 (0.13) | -0.99 (0.13)
  Nasal Congestion Score | -0.19 (0.07) | -0.43 (0.05) | -0.35 (0.06)

15. Secondary Outcome: Change From Baseline in the Individual Symptom Scores Over Period III
Description: as for outcome 13
Time Frame: Baseline, Treatment Period III [Day 2, from drug intake (at 11:00 am) to 3:30 pm]
Population: Only patients with valid individual symptom scores in Period III were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) | Montelukast (MLKT)
Number analyzed (Participants) | 104 | 156 | 151
units on a scale
  Runny Nose Score | -0.52 (0.11) | -1.23 (0.09) | -0.93 (0.09)
  Itchy Nose Score | -0.47 (0.11) | -1.25 (0.09) | -0.89 (0.09)
  Sniffles Score | -0.50 (0.11) | -1.26 (0.09) | -0.96 (0.09)
  Postnasal Drip Score | -0.67 (0.11) | -1.32 (0.09) | -0.97 (0.09)
  Watery Eyes Score | -0.36 (0.11) | -1.11 (0.09) | -0.84 (0.09)
  Itchy Eyes/Ears Score | -0.42 (0.12) | -1.34 (0.10) | -0.87 (0.10)
  Itchy Throat Score | -0.54 (0.11) | -1.15 (0.09) | -0.86 (0.09)
  Cough Score | -0.78 (0.07) | -0.97 (0.06) | -0.84 (0.06)
  Sneezes Score | -0.48 (0.12) | -1.40 (0.10) | -0.78 (0.10)
  Nose Blows Score | -1.22 (0.15) | -2.32 (0.12) | -1.82 (0.13)
  Nasal Congestion Score | -0.43 (0.08) | -0.79 (0.06) | -0.67 (0.07)

16. Secondary Outcome: Change From Baseline in the Individual Symptom Scores Over the Total Treatment Period (Period I + Period II + Period III)
Description: as for outcome 13
Time Frame: Baseline to Day 2
Population: Only patients with valid individual symptom scores during the Total Treatment Period were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) | Montelukast (MLKT)
Number analyzed (Participants) | 105 | 157 | 156
units on a scale
  Runny Nose Score | -0.48 (0.09) | -1.02 (0.07) | -0.84 (0.07)
  Itchy Nose Score | -0.46 (0.09) | -1.05 (0.07) | -0.79 (0.07)
  Sniffles Score | -0.45 (0.09) | -1.05 (0.07) | -0.85 (0.07)
  Postnasal Drip Score | -0.62 (0.09) | -1.11 (0.07) | -0.87 (0.07)
  Watery Eyes Score | -0.44 (0.09) | -0.97 (0.07) | -0.77 (0.07)
  Itchy Eyes/Ears Score | -0.51 (0.10) | -1.17 (0.08) | -0.81 (0.08)
  Itchy Throat Score | -0.54 (0.09) | -1.03 (0.07) | -0.78 (0.07)
  Cough Score | -0.71 (0.06) | -0.86 (0.05) | -0.74 (0.05)
  Sneezes Score | -0.35 (0.10) | -1.23 (0.08) | -0.67 (0.08)
  Nose Blows Score | -1.02 (0.12) | -2.00 (0.10) | -1.58 (0.10)
  Nasal Congestion Score | -0.38 (0.07) | -0.67 (0.05) | -0.61 (0.05)

17. Secondary Outcome: Time to First Feeling of Improvement During Period I
Description: During Period I, the subjects had to record the moment (hh:mm) of first feeling of improvement (compared to Baseline intensity of symptoms).
Time Frame: During Treatment Period 1 [Day 1, from drug intake (at 11:00 am) to 5 hours post-treatment (at 4:00 pm)]
Population: Subjects with no first feeling of improvement were censored at 300 minutes.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) | Montelukast (MLKT)
Number analyzed (Participants) | 66 | 135 | 127
minutes | 101.02 [73.02 to 178.02] | 70.02 [59.02 to 77.02] | 63.02 [60.02 to 73.02]

18. Secondary Outcome: Onset of Action During Period I
Description: The onset of action was defined as the first time point during Period I after initiation of the treatment when the reduction from Baseline in the MSC score for the active treatment group became statistically different from the placebo group and when this significant change was maintained for some period of time.
Time Frame: During Treatment Period 1 [Day 1, from drug intake (at 11:00 am) to 5 hours post-treatment (at 4:00 pm)]
Measure: Number; unit: hours
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) | Montelukast (MLKT)
Number analyzed (Participants) | 105 | 157 | 156
hours | NA — Not applicable for this arm. | 1.5 | 1.5

19. Secondary Outcome: Intensity of Action From Baseline in the MSC Score Over Period I
Description: The intensity of action was measured by the percentage of subjects with categorized percentage change from Baseline in the MSC score over Period I. Categories are defined as following: < 20%, >=20%, < 50%, >=50%, < 70%, >=70% change from Baseline.
Time Frame: Treatment Period 1 [Day 1, from drug intake (at 11:00 am) to 5 hours post-treatment (at 4:00 pm)]
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) | Montelukast (MLKT)
Number analyzed (Participants) | 105 | 157 | 156
percentage of participants
  < 20% | 54.3 | 21.0 | 32.7
  >= 20% | 45.7 | 79.0 | 67.3
  < 50% | 80.0 | 68.8 | 67.9
  >= 50% | 20.0 | 31.2 | 32.1
  < 70% | 95.2 | 87.9 | 92.3
  >= 70% | 4.8 | 12.1 | 7.7

20. Secondary Outcome: Intensity of Action From Baseline in the MSC Score Over Period II
Description: The intensity of action was measured by the percentage of subjects with categorized percentage change from Baseline in the MSC score over Period II. Categories are defined as following: < 20%, >=20%, < 50%, >=50%, < 70%, >=70% change from Baseline.
Time Frame: Treatment Period II [Day 2, from 9:30 am to 11:00 am]
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) | Montelukast (MLKT)
Number analyzed (Participants) | 105 | 157 | 156
percentage of participants
  < 20% | 67.3 | 32.1 | 53.6
  >= 20% | 32.7 | 67.9 | 46.4
  < 50% | 93.3 | 63.5 | 87.4
  >= 50% | 6.7 | 36.5 | 12.6
  < 70% | 98.1 | 83.3 | 95.4
  >= 70% | 1.9 | 16.7 | 4.6

21. Secondary Outcome: Intensity of Action From Baseline in the MSC Score Over Period III
Description: The intensity of action was measured by the percentage of subjects with categorized percentage change from Baseline in the MSC score over Period III. Categories are defined as following: < 20%, >=20%, < 50%, >=50%, < 70%, >=70% change from Baseline.
Time Frame: Treatment Period III [Day 2, from drug intake (at 11:00 am) to 3:30 pm]
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) | Montelukast (MLKT)
Number analyzed (Participants) | 105 | 157 | 156
percentage of participants
  < 20% | 48.1 | 16.7 | 31.8
  >= 20% | 51.9 | 83.3 | 68.2
  < 50% | 84.6 | 48.1 | 63.6
  >= 50% | 15.4 | 51.9 | 36.4
  < 70% | 89.4 | 69.9 | 86.1
  >= 70% | 10.6 | 30.1 | 13.9

22. Secondary Outcome: Variability of Action From Baseline in the MSC Score Over Period I
Description: The variability of action was assessed by the percentage of distribution of the percentage change from Baseline in the MSC score. Categories are defined as following:
  < 20%, 20%-35%, 35%-50%, 50%-65%, 65%-80%, >=80%.
Time Frame: Period 1 [Day 1, from drug intake (at 11:00 am) to 5 hours post-treatment (at 4:00 pm)]
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) | Montelukast (MLKT)
Number analyzed (Participants) | 105 | 157 | 156
percentage of participants
  < 20% | 54.3 | 21.0 | 32.7
  20%-35% | 15.2 | 22.9 | 19.2
  35%-50% | 10.5 | 24.8 | 16.0
  50%-65% | 12.4 | 12.7 | 20.5
  65%-80% | 4.8 | 15.3 | 8.3
  >=80% | 2.9 | 3.2 | 3.2

23. Secondary Outcome: Variability of Action From Baseline in the MSC Score Over Period II
Description: as for outcome 22
Time Frame: Treatment Period II [Day 2, from 9:30 am to 11:00 am]
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) | Montelukast (MLKT)
Number analyzed (Participants) | 105 | 157 | 156
percentage of participants
  < 20% | 67.3 | 32.1 | 53.6
  20%-35% | 17.3 | 19.2 | 16.6
  35%-50% | 8.7 | 12.2 | 17.2
  50%-65% | 3.8 | 17.3 | 6.6
  65%-80% | 1.9 | 10.3 | 3.3
  >=80% | 1.0 | 9.0 | 2.6

24. Secondary Outcome: Variability of Action From Baseline in the MSC Score Over Period III
Description: as for outcome 22
Time Frame: Treatment Period III [Day 2, from drug intake (at 11:00 am) to 3:30 pm]
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) | Montelukast (MLKT)
Number analyzed (Participants) | 105 | 157 | 156
percentage of participants
  < 20% | 48.1 | 16.7 | 31.8
  20%-35% | 21.2 | 17.9 | 14.6
  35%-50% | 15.4 | 13.5 | 17.2
  50%-65% | 3.8 | 14.1 | 17.2
  65%-80% | 8.7 | 17.9 | 14.6
  >=80% | 2.9 | 19.9 | 4.6

25. Secondary Outcome: Global Satisfaction of the Subjects at the End of Period III
Description: Global satisfaction was evaluated at the end of Period III by the subject on a Visual Analog Scale (VAS) ranging from 0 (very dissatisfied) to 100 mm (very satisfied).
Time Frame: At the end of Period III (Day 2)
Population: Only subjects with valid data for Global Satisfaction (VAS Score) were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) | Montelukast (MLKT)
Number analyzed (Participants) | 104 | 156 | 152
units on a scale | 32.42 (31.05) | 53.94 (32.95) | 41.80 (32.10)

26. Secondary Outcome: Percentage of Subjects, at the End of Period III Who Are Willing to Take the Same Medication During the Next Pollen Season
Description: At the end of Period III, each subject without reference to the Symptom Diary Card (SDC) answered to the question: "Do you want to take the same treatment during the next pollen season?" (yes or no).
Time Frame: At the end of Period III (Day 2)
Population: Only subjects with valid data were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) | Montelukast (MLKT)
Number analyzed (Participants) | 104 | 156 | 152
percentage of participants | 23.1 | 49.4 | 32.9

ADVERSE EVENTS:
Time Frame: Adverse events were recorded in Study Phase II and in Study Phase III (Day 1 and Day 2), before and after each pollen exposure.
Description: Adverse Events refer to the Safety Population consisting of all subjects who were dispensed medication.
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) | Montelukast (MLKT)
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/157 | 0/156
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/157 | 0/156
Other Adverse Events (participants affected / at risk) | 9/105 | 13/157 | 18/156
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (PBO) (N=105) | Levocetirizine (LCTZ) (N=157) | Montelukast (MLKT) (N=156)
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 1 | 0
Eye swelling (Eye disorders) | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 3
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 2 | 0
Feeling hot (General disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0
Body temperature increased (Investigations) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Nodule on extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 5
Sinus headache (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 2 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 3
Urticaria localised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days